CLINICAL TRIAL: NCT06636266
Title: Examining Scottish Chiropractic Professional Identity Using Chiropractic Professional Identity Scales
Acronym: PI_Chiro
Status: Recruiting | Type: Observational
Sponsor: Scotland College of Chiropractic (Other)
Responsible Party: Principal Investigator, Alice Cade, Senior lecturer and research fellow, Scotland College of Chiropractic
Other Study IDs: 348918
Record Dates: First submitted 2024-09-12; First posted 2024-10-10 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Professional Identity Formation
Keywords: Student; identity
MeSH Terms: conditions — Social Identification

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chiropractors: Practising in Scotland at the time of the survey/study
  Interventions: Other: Survey using a questionnaire.
- Chiropractic students: Enrolled in the Scotland College of Chiropractic at the time of the study
  Interventions: Other: Survey using a questionnaire.

INTERVENTIONS:
Other: Survey using a questionnaire. — This research will examine any potential differences in the professional identity of Scottish chiropractors utilising the Chiropractic Professional Identity Embodiment Scale (CPIES) and the Subtype Orientation Scale (CPISOS).

SUMMARY:
This research will examine any potential differences in the professional identity of Scottish chiropractors utilising the Chiropractic Professional Identity Embodiment Scale (CPIES) and the Subtype Orientation Scale (CPISOS). Data will be collected through an online web-based survey. Potential statistical relationships with variables such as age, gender, ethnicity, and previous education on chiropractic professional identity (CPI) will also be explored. This study expands upon prior investigations to further explore the CPI of chiropractic identity internationally. Additionally, the data gleaned from this study could be used as a platform to build understanding and interprofessional relationships within Scotland and, potentially, to aid in working towards greater recognition of chiropractic within Spain. This research could assist Scottish chiropractors in creating better avenues to strengthen their professional identity to help future chiropractors thrive in Europe.

DETAILED DESCRIPTION:
Research Question(s) Using the CPIES and CPISOS, does the strength of chiropractic professional identity (CPI) vary across Scottish chiropractors? For the CPIES and CPISOS, are there any influences on CPI across age, gender, ethnicity, or pre-professional educational variables?

Rationale and Significance of the Study By aiming to understand CPI and its drivers, the investigators may be able to strengthen and develop chiropractors' professional identity without homogenisation. A strong professional identity facilitates the taking up of professional responsibilities, promotes a sense of belonging and professional socialisation, increases competence, fosters greater belonging, stability, and esteem, and promotes enhanced decision-making and confidence. These have been shown to enhance trust and patient safety and ultimately lead to better practice and patient outcomes. By better understanding CPI, and through the use of the Chiropractic Professional Identity Embodiment Scale (CPIES) and the Subtype Orientation Scale (CPISOS), the investigators may be able to identify potential divisions or areas of friction in chiropractic curriculum and to better support the profession.

Chiropractic research has shown that burnout and professional dissatisfaction may be a consequence of poor professional identity. In a sample of chiropractors, the CPIES and CPISOS may help to identify areas of professional identity that could be strengthened, and that may ultimately improve professional satisfaction and success.

This project will also allow us to collect demographic data of Scottish chiropractors, which may also assist in understanding the profession in greater detail and depth.

Literature/Past Research Review

Simply belonging to a profession does not alone determine one's professional identity; rather, variation exists in beliefs relating to one's occupation. 11 While chiropractic is an established health profession, there is a lack of clarity about the role of chiropractic in healthcare. There is disagreement on what characterises the chiropractic profession, its philosophy, and scope of practice. Chiropractors themselves have reported being challenged at times by the unclear public identity of the profession brought about by contrasting practice styles.

Studies exist on chiropractors' attitudes and beliefs on professional identity. In North America, New Zealand, and Australia, pre-chiropractic education and the geographic region have been shown to be associated with differences in professional identity. In North America, chiropractic students report a preference for participating in mainstream health care and a desire to hold to traditional chiropractic theories and practices, being elements of various domains of chiropractic professional identity. Professional identity has been said to begin with formal education and has been researched with undergraduate chiropractic students. Common themes of an interplay between professional association membership status, pre-chiropractic education, and institutional philosophy have been cited as being determining factors in identity construction.

Limitations of these current studies exist, the main being that the surveys employed in the research were not psychometrically validated. Additionally, the surveys differed in each study, making generalisability and comparisons difficult. These issues may be remedied through the use of a consistent psychometrically robust scale such as the CPIES. The CPIES was derived through mixed methods research using a qualitative phase that used one-to-one cognitive interviews of 15 expert key informants to inform and develop a pool of 92-candidate items across six known CPI domains. These items were then tested on 231-participants (New Zealand chiropractors and chiropractic students) for psychometric robustness. The final CPIES comprised 22-items and was found to be a valid and reliable measure of CPI. It has been identified that further research is needed to improve the understanding of measurement properties of tools used in research and to aid their selection and use. 25, and this research aims to begin to fill some of these gaps in knowledge.

Primary research question: Using the Chiropractic Professional Identity Embodiment Scale (CPIES) and Subtype Orientation Scale (CPISOS), does the strength of chiropractic professional identity (CPI) vary across Scottish chiropractors?

Secondary research question: For the Chiropractic Professional Identity Embodiment Scale (CPIES) and Subtype Orientation Scale (CPISOS), are there any influences on chiropractic professional identity (CPI) across age, gender, ethnicity, or pre-professional educational variables?

Design of the Study

Study design and setting

This research is quantitative descriptive study to analyse CPIES and CPISOS questionnaire data across Scottish chiropractors and chiropractic students. The study will be conducted primarily at the Scotland College of Chiropractic. The lead investigator for the project is Dr Alice Cade.

Participants

All practising Scottish chiropractors and currently enrolled chiropractic students will be invited to take part in this study. Potential participants will not be eligible if they are practising outside of Scotland or enrolled to study chiropractic in an institute outside of Scotland.

Procedure

Participants will be asked to review the purpose of this study and the participant selection criteria, indicate their agreement to participate, and complete an online web-based survey to rate their beliefs towards 22-CPIES and 21-CPISOS statements and one CPI self-categorisation question on a 5-point Likert scale. The survey is anticipated to take 10 minutes to complete. Data will be anonymous and collected on a platform such as Qualtrics to be analysed by R software.

The sample size was based on calculations recommended by Bartlett (2001), where the alpha level a priori at .05, and based on a five-point scale, the level of acceptable error at 3%, and estimated the standard deviation of the scale was 1.25. As the sample size calculated exceeded 5% of the possible population, the available sample size was corrected using Cochran's (1977) formula, resulting in a recommended sample size of 78.

There are approximately 90 practising chiropractors and 26 students enrolled at the Scotland College of Chiropractic, and the investigators hope to gain a response from over half of these potential participants, which previous studies have found achievable.

Statistical analyses

Primary outcomes: A unidimensional score and six sub-scale numerical scores from the Chiropractic Professional Identity Embodiment Scale (CPIES).

Secondary outcomes: A unidimensional measurement of chiropractic practitioner subtypes numerical score from the Chiropractic Professional Identity Subtype Orientation Scale (CPISOS).

A numerical score from the self-categorisation of chiropractors' professional identity along a philosophical continuum scale.

Demographical details will be analysed through descriptive statistics. Pragmatic use of additional statistical analyses between year groups for the CPIES and CPISOS will be used, and various correlations will be investigated for subscale and sum scores.

Location The data will be collected online, and the research will be hosted by the Scotland College of Chiropractic.

ELIGIBILITY:
Inclusion Criteria:

* All practising Scottish chiropractors and currently enrolled chiropractic students will be invited to participate in this study.

Exclusion Criteria:

* Potential participants will not be eligible if they are practising outside of Scotland or enrolled to study chiropractic in an institute outside of Scotland.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All practising Scottish chiropractors and currently enrolled chiropractic students will be invited to participate in this study. Potential participants will not be eligible if they are practising outside of Scotland or enrolled to study chiropractic in an institute outside of Scotland.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2024-10-20 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Chiropractic Professional Identity Embodiment Scale | Baseline
  A unidimensional score and six sub-scale numerical scores from the Chiropractic Professional Identity Embodiment Scale (CPIES). There are 15 questions, and each question is measured by a 5 point likert scale ranging from "strongly Disagree" (1) to "Strongly Agree" (5). The minimum value is 15 maximum value is 75. A lower/higher score does not denote an better or worse outcome, but places the participant, with further weighted analyses (see here for review: https://www.sciencedirect.com/science/article/pii/S1744388124000136#sec2) into a category of practitioner: Traditional, centrist, or musculoskeletal focussed. The six subscales measure participants responses in 6 subscales: Chiropractic History, Engagement & Interactions, Ethics & Standards of Practice, Philosophy & Motivations, Pride & Attitude, Pride & Attitude.

SECONDARY OUTCOMES:
Chiropractic Professional Identity Subtype Orientation Scale (CPISOS). | Baseline
  A unidimensional measurement of chiropractic practitioner subtypes numerical score from the Chiropractic Professional Identity Subtype Orientation Scale (CPISOS).
  There are 19 questions, and each question is measured by a 5 point likert scale ranging from "strongly Disagree" (1) to "Strongly Agree" (5). The minimum value is 19 maximum value is 95. A lower/higher score does not denote a better or worse outcome, but places the participant, with further weighted analyses, into the type of chiropractic they practise, as opposed to the Chiropractic Professional Identity Embodiment Scale (CPIES) which categories the professional identity based on what the chiropractor believes about themselves and their own identity.
Chiropractic philosophical continuum scale | Baseline
  A numerical score from the self-categorisation of chiropractors' professional identity along a philosophical continuum scale.
  This is a 5 question survey with Yes/No answers possible. The combination of responses places the practitioner in one of three possible identities
  1. = I am fundamentally a Vertebral Subluxation (VS, meaning traditional) focused chiropractor.
  2. = I am fundamentally a Musculoskeletal (MSK) focused chiropractor.
  3. = I am fundamentally a centrist (shared aspects of VS and MSK treatment focused chiropractic) chiropractor.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Cade, PhD, Principal Investigator — New Zealand College of Chiropractic
Locations (1):
- Scotland College of Chiropractic, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The IPD will be available on reasonable request to the chief investigators by other researchers